CLINICAL TRIAL: NCT04869592
Title: Phase I/II Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Recombinant SARS-CoV-2 Vaccine (CHO Cell) in Healthy People Aged 3 Years and Older
Brief Title: A Clinical Trial to Evaluate the Recombinant SARS-CoV-2 Vaccine (CHO Cell) for COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Zhong Sheng Heng Yi Pharmaceutical Technology Co., Ltd. (Unknown); Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-YM-006-02
Record Dates: First submitted 2021-04-24; First posted 2021-05-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Phase 1 low-dose group (Experimental)
  Interventions: Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 1 high-dose group (Experimental)
  Interventions: Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 1 placebo group (Placebo Comparator)
  Interventions: Biological: placebo
- Phase 2 low-dose group A (Experimental)
  Interventions: Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 low-dose group B (Experimental)
  Interventions: Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 low-dose group C (Experimental)
  Interventions: Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 low-dose group D (Experimental)
  Interventions: Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 high-dose group A (Experimental)
  Interventions: Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 high-dose group B (Experimental)
  Interventions: Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 high-dose group C (Experimental)
  Interventions: Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 high-dose group D (Experimental)
  Interventions: Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell)
- Phase 2 placebo group A (Placebo Comparator)
  Interventions: Biological: placebo
- Phase 2 placebo group B (Placebo Comparator)
  Interventions: Biological: placebo
- Phase 2 placebo group C (Placebo Comparator)
  Interventions: Biological: placebo
- Phase 2 placebo group D (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell) — Intramuscular injection of low-dose Recombinant SARS-CoV-2 Vaccine (CHO cell) in the deltoid muscle of the upper arm
  Arms: Phase 1 low-dose group; Phase 2 low-dose group A; Phase 2 low-dose group B; Phase 2 low-dose group C; Phase 2 low-dose group D
Biological: high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell) — Intramuscular injection of high-dose Recombinant SARS-CoV-2 Vaccine (CHO cell) in the deltoid muscle of the upper arm
  Arms: Phase 1 high-dose group; Phase 2 high-dose group A; Phase 2 high-dose group B; Phase 2 high-dose group C; Phase 2 high-dose group D
Biological: placebo — Intramuscular injection of placebo in the deltoid muscle of the upper arm
  Arms: Phase 1 placebo group; Phase 2 placebo group A; Phase 2 placebo group B; Phase 2 placebo group C; Phase 2 placebo group D

SUMMARY:
phase I study will evaluate safety and immunogenicity of a recombinant SARS-CoV-2 vaccine (CHO cell) in Chinese healthy population aged 3 years and older. 300 subjects will be enrolled and divided into 5 age groups: 18-59 years old group, 60-69 years old group, ≥70 years old group, 9-17 years old group and 3-8 years old group. In each group, there are two regimen cohort: low-dose at 0,30, 60 schedule and high-dose at 0,30,60 schedule. The subjects in regimen cohort will be randomized to receive vaccines or placebos at a ratio of 2:1.

Phase II clinical study will explore dose and immunization procedures in 5 age groups, including 18-59 years old group, 60-69 years old group, ≥70 years old group, 9-17 years old group, and 3-8 years old group, with a total of 3280 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age range: healthy people aged 3 years and and older who can provide legal identification;
* The subject and/or his legal guardian and/or his entrusted person can understand the study procedures and informed consent, voluntarily sign informed consent form, and be able to comply with the requirements of the clinical study protocol;
* Inquired about medical history and physical examination, the investigator judged that the health condition is good;
* No history of SARS-CoV-2 vaccination before enrollment;
* Females of childbearing age (menarche to menopause) are not pregnant at the time of enrollment (negative urine pregnancy test), not breastfeeding, and have no birth plan within 12 months after enrollment; effective contraception will be taken within 2 weeks before enrollment;
* During the entire study follow-up period, be able and willing to complete the entire prescribed study plan.

Exclusion Criteria:

First Dose Exclusion Criteria：

* Confirmed cases of SARS-CoV-2 infection, suspected cases, asymptomatic infections, or close contacts with the above population (check "China Disease Prevention and Control Information System");
* Axillary body temperature is not less than 37.3℃ (older than 14 years) before vaccination, and axillary body temperature is not less than 37.5℃ (14 years or younger) before vaccination;
* Positive in SARS-CoV-2 IgG and IgM antibody screening;
* Have a history of SARS virus infection (self-report, on-site inquiry);
* Fever (axillary temperature is not less than 37.3℃), dry cough, fatigue, nasal, congestion, runny nose, sore throat, myalgia, diarrhea, shortness of breath, or dyspnea within 14 days before vaccination;
* Before vaccination, the results of blood biochemistry, blood routine, urine routine, and coagulation function related indexes are abnormal, which exceed the reference value range, and have clinical significance abnormalities (only refers to phase I);
* Previous severe allergic reaction to vaccination (such as acute allergic reaction, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain);
* Allergic to any component of the study vaccine (such as aluminum, histidine, etc.);
* Have a history of convulsions, epilepsy, encephalopathy, long-term alcoholism and drug abuse, thyroidectomy, infectious diseases, mental illness or family history;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Known or suspected diseases include: severe respiratory disease, severe liver and kidney disease, severe cardiovascular disease, drug-uncontrollable hypertension (systolic blood pressure is not less than 140mmHg, diastolic blood pressure is not less than 90mmHg), high blood glucose, diabetic complications , Malignant tumors, various acute diseases or acute attacks of chronic diseases;
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* Have a history of abnormal coagulation function (such as coagulation factor deficiency, coagulopathy);
* Asthenia or splenectomy, functional asthenia caused by any situation;
* Are receiving anti-TB (tuberculosis) treatment;
* Have received immune enhancement or inhibitor therapy within 3 months (continuous oral or instillation for more than 14 days);
* Have received a live attenuated vaccine within 28 days before vaccination, or received other vaccines within 14 days before vaccination;
* Have received blood products within 3 months before vaccination;
* Have received other study drugs within 6 months before vaccination;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* Other conditions considered by the investigator to be inappropriate for participation in the study.

Exclusion criteria for the second and third doses of vaccination

* Positive urine pregnancy test;
* Have a high fever (axillary temperature is not less than 39.0℃) for three days and severe allergic reaction after the previous dose of vaccination;
* Severe adverse reactions that are causally related to the previous dose of vaccination;
* For those newly discovered or newly identified after the previous dose of vaccine that does not meet the first dose selection criteria or meets the first dose exclusion criteria, the investigator will determine whether to continue participating in the study;
* Other exclusion reasons considered by the investigator.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3100 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
the incidence and severity of any adverse reactions/events within 30 minutes after each dose of vaccination | through 30 minutes after each dose
  Phase 1
the incidence of abnormal blood biochemistry, blood routine, blood coagulation function and urine routine on the 4th day after each dose of vaccination | 4th day each dose
  Phase 1
the incidence and severity of adverse reactions/events within 0-7 days after each dose of vaccination | through 7 days after each dose
  Phase 1
the incidence and severity of non-collective adverse reactions/events within 30 days after each dose of vaccination | through 30 days after each dose
  Phase 1
the incidence and severity of adverse events leading to withdrawal within 30 days after each dose of vaccination | through 30 days after each dose
  Phase 1
the incidence of SAE from the first dose of vaccination to 12 months after the full course of vaccination | up to 12 months after the full course of vaccination
  Phase 1
the incidence of AESI from the first dose of vaccination to 12 months after the full course of vaccination | up to 12 months after the full course of vaccination
  Phase 1
Geometric mean Titer of SARS-CoV-2 specific neutralizing antibody(wild Strains) on the 15th day after the full course of vaccination | 15th day after the full course of vaccination
  Phase 1
the incidence and severity of any adverse reactions/events within 30 minutes after each dose of vaccination | through 30 minutes after each dose
  Phase 2
the incidence and severity of adverse reactions/events within 0-7 days after each dose of vaccination | through 7 days after each dose
  Phase 2
the incidence and severity of non-collective adverse reactions/events within 30 days after each dose of vaccination | through 30 days after each dose
  Phase 2
the incidence and severity of non-collective adverse reactions/events within 40 days after each dose of vaccination | through 40 days after each dose
  Phase 2
the incidence and severity of non-collective adverse reactions/events within 60 days after each dose of vaccination | through 60 days after each dose
  Phase 2
the incidence and severity of adverse events leading to withdrawal within 30 days after each dose of vaccination | through 30 days after each dose
  Phase 2
the incidence and severity of adverse events leading to withdrawal within 40 days after each dose of vaccination | through 40 days after each dose
  Phase 2
the incidence and severity of adverse events leading to withdrawal within 60 days after each dose of vaccination | through 60 days after each dose
  Phase 2
the incidence of SAE from the first dose of vaccination to 12 months after the full course of vaccination | up to 12 months after the full course of vaccination
  Phase 2
the incidence of AESI from the the first dose of vaccination to 12 months after the full course of vaccination | up to 12 months after the full course of vaccination
  Phase 2
Geometric mean Titer of SARS-CoV-2 specific neutralizing antibody (wild Strains) on the 15th day after the full course of vaccination | 15th day after the full course of vaccination
  Phase 2

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (Live SARS-CoV-2 neutralization assay) On the 30th day after the full course of vaccination, the neutralizing antibody level (wild Strains) | 30th day after the full course of vaccination
  Phase 1
Seroconversion and Geometric Mean Titer (GMT) of SARS-CoV-2-Specific Binding Antibody (IgG) Before each dose, the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after full course of vaccination | before each dose , the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 1
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (Pseudovirus neutralization assay) in the 18-59 years old group before each dose and on the 15th and 30th day after the full course of vaccination | before each dose，the 15th, 30th day after the full course of vaccination
  Phase 1
Geometric Mean Titer (GMT) of SARS-COV-2 specific neutralizing antibody (live SARS-CoV-2 neutralization assay)) On the 30th day after the full course of vaccination | 30th day after the full course of vaccination
  Phase 2
Two-dose group: the neutralizing antibody levels (live SARS-CoV-2 neutralization assay) before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Two-dose group: Seroconversion before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Two-dose group: Binding Antibody (IgG) before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Three-dose group: the neutralizing antibody levels (live SARS-CoV-2 neutralization assay) before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Three-dose group:Seroconversion before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Three-dose group:Binding Antibody (IgG) before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination | before each dose，the 15th day after the second dose, the 15th, 30th, 90th, 180th, 360th day after the full course of vaccination
  Phase 2
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (Pseudovirus neutralization assay) in the 18-59 years old 0,30,60 group before each dose , the 15th and 30th day after the full course of vaccination | before each dose, 15th, 30th day after the full course of vaccination
  Phase 2

CONTACTS AND LOCATIONS:
Locations (1):
- Ning ling Center for Disease Control and Prevention, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: No